CLINICAL TRIAL: NCT07253831
Title: Effect of Hand Reflexology Massage on Fatigue and Anxiety Level Among Patients Undergoing Hemodialysis: a Randomized Control Trial.
Brief Title: Effect of Hand Reflexology Massage on Fatigue and Anxiety Among Patients Undergoing Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Sabah Kareem Jabbar Alwan, Master's Student / Principal Investigator, Kufa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKJ-HRM-HD-2025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: End Stage Kidney Disease (ESRD); Hemodialysis; Anxiety; Fatigue; Reflexology
Keywords: Psychological distress; Quality of life; Renal failure; Randomized controlled trial; Nursing intervention; Complementary therapy; Hemodialysis; Fatigue; Anxiety; Non-pharmacological intervention; Hand Reflexology Massage; Reflexology
MeSH Terms: conditions — Kidney Failure, Chronic; Anxiety Disorders; Fatigue; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: This is a two-arm, assessor-blinded, randomized controlled trial. Participants are randomly assigned to either receive hand reflexology massage in addition to routine care or to continue with routine care alone.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Reflexology Massage (Experimental): Participants in this group will receive standard hemodialysis care plus eight sessions of hand reflexology massage over four weeks. Each session, lasting approximately 27 minutes, will be conducted twice a week during their dialysis treatment and will focus on specific reflex points (solar plexus, diaphragm line, adrenal glands, kidneys, pituitary gland, and heart point on the left hand) to promote relaxation and reduce fatigue and anxiety.
  Interventions: Procedure: Hand Reflexology Massage
- Standard Care (Active Comparator): Participants in this group will receive routine hemodialysis care only, without any additional hand reflexology massage. This includes standard nursing care, monitoring, and medical management as per the center's protocol. This group serves as a control to compare against the intervention group receiving hand reflexology.
  Interventions: Procedure: Standard

INTERVENTIONS:
Procedure: Hand Reflexology Massage — The intervention is a standardized Hand Reflexology Massage (HRM) for adults on maintenance hemodialysis, applied twice weekly for four weeks during dialysis. Each 27-minute session follows a structured three-phase protocol: 7 minutes of preparatory relaxation, 18 minutes of targeted stimulation of key reflex points (Solar Plexus, Diaphragm, Adrenal/Kidney, Pituitary, and Heart on the left hand), and 2 minutes of concluding relaxation. Pressure is applied systematically using thumb or index finger. Male patients are treated by the principal investigator, females by a trained female co-researcher. This evidence-based, non-invasive therapy differs from general hand massage by focusing on validated reflex points, reducing fatigue and anxiety, and integrating safely into dialysis care.
  Arms: Hand Reflexology Massage
Procedure: Standard — The control group receives standard care, which consists of routine hemodialysis treatment and standard nursing care as per the established protocols at Fatima Al-Zahraa and Al-Hayat Hemodialysis Centers. This includes monitoring vital signs, managing dialysis parameters, administering prescribed medications, providing general health education, and offering emotional support during the treatment sessions.
  Arms: Standard Care

SUMMARY:
The goal of this clinical trial is to learn if hand reflexology massage can help reduce fatigue and anxiety in adult patients undergoing hemodialysis treatment. The main questions it aims to answer are:

* What are the levels of fatigue and anxiety in hemodialysis patients?
* Is hand reflexology massage more effective than usual care in reducing fatigue and anxiety after eight sessions?
* Do these improvements last over time?
* Does a patient's age, gender, education level, how long they've been on dialysis, or their financial status affect how much they benefit from the massage?

Researchers will compare patients who receive hand reflexology massage plus standard care to those who receive only standard care to see if the massage leads to greater reductions in fatigue and anxiety.

Participants will:

* Be randomly assigned to one group that receives hand reflexology massage or another group that continues with routine care only
* Attend 8 short sessions (about 27 minutes each) of hand reflexology massage over four weeks, given during their regular dialysis visits
* Complete brief questionnaires about their fatigue and anxiety levels before the study starts, after the 4th session, and after the 8th session
* Continue their normal medical treatments throughout the study

This study focuses on a safe, non-drug therapy that nurses can easily provide. Hand reflexology involves gentle pressure on specific points of the hands linked to stress relief and relaxation. It is chosen because it is practical during dialysis, avoids touching swollen or sensitive feet, and respects cultural preferences. The results could help improve the comfort and well-being of hemodialysis patients in Iraq and similar healthcare settings.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) designed to evaluate the effectiveness of Hand Reflexology Massage (HRM) in reducing fatigue and anxiety levels among adult patients undergoing maintenance hemodialysis at Fatima Al-Zahraa and Al-Hayat Hemodialysis Centers in Al-Diwaniyah, Iraq. The research addresses a critical need, as patients with End-Stage Renal Disease (ESRD) on hemodialysis often suffer from debilitating symptoms like severe fatigue-reported in 60-97% of cases-and high rates of anxiety, which significantly impair their quality of life. Standard pharmacological treatments are often limited for these patients due to altered drug metabolism and potential side effects, making safe, non-drug therapies an important area of investigation.

The study will enroll 104 participants who meet specific criteria, including being over 18 years old, having been on hemodialysis for at least three months, and experiencing measurable levels of fatigue and anxiety. Participants will be randomly assigned to one of two groups: an intervention group that receives standard care plus eight sessions of HRM, or a control group that receives only standard care. The HRM protocol is based on established reflexology principles and adapted from previous clinical studies. Each session will last approximately 27 minutes and will be conducted twice a week over four weeks during the patients' regular dialysis appointments.

The HRM technique involves a structured sequence of movements performed on both hands. It begins with preparatory relaxation techniques such as the "Butterfly Touch" and "Phoenix Rising," followed by focused stimulation of key reflex points believed to influence stress and well-being. These include the solar plexus (for emotional calm), the diaphragm line (to support breathing), the adrenal glands and kidneys (to help manage the body's stress response and fatigue), the pituitary gland (for hormonal balance), and the heart point on the left hand (for emotional health). The procedure was standardized to ensure consistency, with male participants treated by the principal researcher and female participants treated by a trained female co-researcher to respect cultural norms.

The primary goal is to measure changes in fatigue and anxiety levels. Fatigue will be assessed using the Arabic version of the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F), a validated 13-item questionnaire. Anxiety will be measured using the Arabic version of the Beck Anxiety Inventory (Ar-BAI), a 21-item self-report scale. Data will be collected at three time points: before the intervention begins (T₀), after the fourth session (T₁), and after the eighth and final session (T₂). This allows researchers to observe not only the immediate effects but also any cumulative benefits of the therapy.

The study is grounded in Roy's Adaptation Model, a nursing theory that views patients as adaptive systems responding to environmental stressors. In this context, chronic illness and hemodialysis are the primary stressors, while HRM is introduced as a therapeutic intervention to promote physiological and psychological adaptation. By potentially stimulating the parasympathetic nervous system and promoting relaxation, HRM may help patients better adapt to the challenges of their condition.

This research is significant because, despite evidence supporting foot reflexology, no rigorous RCT has specifically examined the combined effect of HRM on both fatigue and anxiety in Iraqi hemodialysis patients. The findings could provide strong evidence for a simple, cost-effective, and culturally appropriate nursing intervention that can be easily integrated into routine care. If effective, HRM could empower nurses to improve patient comfort and well-being, reduce reliance on medication, and enhance the overall quality of care in resource-limited settings like Iraq.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Diagnosed with End-Stage Renal Disease (ESRD) and undergoing maintenance hemodialysis for at least three months.
* Receiving hemodialysis treatment two or three times per week.
* Fully alert, conscious, and able to communicate clearly.
* Able to understand the Arabic language.
* Demonstrates measurable levels of fatigue as assessed by the FACIT-Fatigue Scale.
* Demonstrates measurable levels of anxiety as assessed by the Beck Anxiety Inventory (Ar-BAI).
* Willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Presence of ulcers, wounds, burns, infections, or skin diseases on the hands or forearms.
* Deformities, fractures, or orthopedic disorders affecting the hands or upper limbs.
* Peripheral neuropathy, vascular problems, or Raynaud's phenomenon in the hands.
* Diagnosis of major psychiatric disorders (e.g., psychosis, bipolar disorder, generalized anxiety disorder).
* Active systemic diseases that contribute to fatigue or anxiety (e.g., cancer, heart failure, lupus).
* Use of sedatives, anxiolytics, or sleeping pills within 48-72 hours prior to data collection.
* Current use of complementary or alternative therapies aimed at managing anxiety or fatigue.
* History of drug or alcohol abuse.
* Presence of implanted cardiac devices (e.g., pacemaker, implantable cardioverter defibrillator).
* Hemodynamic instability or unstable vital signs during hemodialysis sessions.
* Refusal or inability to complete the required reflexology sessions or study questionnaires.
* Missing more than two scheduled intervention sessions during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue Levels as Measured by the Arabic FACIT-Fatigue Scale (FACIT-F) | 4 weeks
  The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F, Version 4) is a validated 13-item questionnaire used to assess fatigue severity and its impact on quality of life over the past week. Each item is scored on a 5-point Likert scale (0 = "Not at all" to 4 = "Very much"). After reverse-scoring specific items, the total score ranges from 0 to 52, with higher scores indicating lower levels of fatigue. This measure will be administered to participants in both the intervention and control groups at three time points to evaluate the effect of Hand Reflexology Massage.
Change in Anxiety Levels as Measured by the Arabic Beck Anxiety Inventory (Ar-BAI) | 4 weeks
  The Arabic version of the Beck Anxiety Inventory (Ar-BAI) is a 21-item self-report scale used to measure the severity of anxiety symptoms experienced in the past week. Each item is scored from 0 ("Not at all") to 3 ("Severely-it bothered me a lot"), resulting in a total score ranging from 0 to 63. Higher scores indicate greater anxiety severity. This measure will be used to compare changes in anxiety between the two study groups across the same three assessment periods.

IPD SHARING:
Plan to Share IPD: No
The study does not plan to share Individual Participant Data (IPD) due to the sensitive nature of the data collected, which includes personal health information from a vulnerable patient population undergoing hemodialysis in Iraq. The informed consent obtained from participants did not include provisions for data sharing beyond the research team, and the ethical approval from the University of Kufa's Medical Ethical Committee restricts the dissemination of raw data to protect participant confidentiality and comply with local data protection regulations. Additionally, the small sample size and the specific cultural context of the study limit the generalizability of the data, making it unsuitable for secondary analysis by external researchers.

REFERENCES:
- [Result] Heidari, F., Rejeh, N., Heravi-Karimooi, M., Tadrisi, S. D., & Vaismoradi, M. (2017). Effect of short-term hand reflexology on anxiety in patients before coronary angiography: A randomized placebo controlled trial. European Journal of Integrative Medicine, 16, 1-7. https://doi.org/10.1016/j.eujim.2017.09.010
- [Result] Ali EA, Awad WHA, Khedr MA, Rabie EAEGA. Effect of hand reflexology in ameliorating anxiety, pain, and fatigue among patients undergoing coronary angiography. BMC Complement Med Ther. 2023 Nov 24;23(1):425. doi: 10.1186/s12906-023-04256-6. PMID 38001461
- [Result] Rejeh N, Tadrisi SD, Yazdani S, Saatchi K, Vaismoradi M. The Effect of Hand Reflexology Massage on Pain and Fatigue in Patients after Coronary Angiography: A Randomized Controlled Clinical Trial. Nurs Res Pract. 2020 Aug 29;2020:8386167. doi: 10.1155/2020/8386167. eCollection 2020. PMID 32908698